CLINICAL TRIAL: NCT03796598
Title: Fecal Microbiota Transplant in Veterans With Cirrhosis
Brief Title: FMT in Cirrhosis and Hepatic Encephalopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: GAST-001-18S; CX001076 (Other Grant/Funding Number: Office of Research and Development, VA)
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
Keywords: fecal microbial transplant; cirrhosis; hepatic encephalopathy
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into 4 groups via randomization
  Group 1: Dual oral and rectal FMT, Group 2: Oral FMT and rectal placebo, Group 3: Oral placebo and rectal FMT and Group 4: Oral and rectal placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Oral and rectal placebo at visit 2 Oral placebo at day 30
  Interventions: Other: Placebo
- Group 3: Oral placebo and rectal FMT (Active Comparator): Oral placebo and rectal FMT at visit 2 Oral placebo at day 30
  Interventions: Drug: Fecal Microbial Transplant Enema; Other: Placebo
- Group 2: Oral FMT and rectal placebo (Active Comparator): Oral FMT and rectal placebo at visit 2 Oral FMT at day 30
  Interventions: Drug: Fecal Microbial transplant Capsules
- Group 1: Dual Oral and rectal FMT (Experimental): Dual Oral and rectal FMT at visit 2 Oral FMT at day 30
  Interventions: Drug: Fecal Microbial transplant Capsules; Drug: Fecal Microbial Transplant Enema

INTERVENTIONS:
Drug: Fecal Microbial transplant Capsules — Oral capsules of FMT
  Arms: Group 1: Dual Oral and rectal FMT; Group 2: Oral FMT and rectal placebo
Drug: Fecal Microbial Transplant Enema — FMT enema
  Arms: Group 1: Dual Oral and rectal FMT; Group 3: Oral placebo and rectal FMT
Other: Placebo — Placebo
  Arms: Group 3: Oral placebo and rectal FMT; Placebo

SUMMARY:
Patients with end stage of liver disease or cirrhosis can develop confusion due to high ammonia and inflammation. This confusion is brought upon by changes in the bacteria in the bowels and may not respond to current standard of care treatments. Repeated episodes of confusion can make it difficult for patients to function and may result in multiple admissions to the hospital and burden on the family. The investigators have studied using a healthy person's stool to replace the bowel bacteria, called fecal microbial transplant, in small studies with good results. In this trial the investigators propose to perform these procedures using an upper and lower route in Veterans who suffer from this condition and follow them for safety and HE and related hospitalizations over 6 months. The investigators will compare this to placebo treatments and hope that this intervention can improve the health and daily functioning of affected patients.

DETAILED DESCRIPTION:
Indication: Cirrhosis and hepatic encephalopathy

Study Objectives: To evaluate the safety and tolerability of fecal transplant in patients with cirrhosis and hepatic encephalopathy

Rationale and Supporting Evidence:

Hepatic encephalopathy affects 30-45% of patients with cirrhosis and adversely affects survival in these patients. The mainstay of treatment for hepatic encephalopathy (HE) has long been the manipulation of the gut flora through antibiotics, prebiotics or probiotics. The current first and second line therapies for HE in the US are lactulose and rifaximin respectively that uniquely act within the confines of the gut lumen with encouraging clinical results. However, there is a subset of patients with HE that continues to recur despite being on both treatments. This patient group is at a higher risk of poor outcomes because HE has now been removed from liver transplant priority and multiple episodes of HE can result in cumulative brain injury which may be irreversible. Therefore, the prevention of recurrent HE is an important therapeutic goal.

The investigators' group and other reports have shown that patients with HE and cirrhosis are more likely to have overgrowth of potentially pathogenic bacterial taxa such as Enterobacteriaceae and reduction of autochthonous species such as Lachnospiraceae and Ruminococcaceae in the stool and the colonic mucosa. This has been linked to poor performance on cognitive tests that are a hallmark of HE and with increased systemic inflammation in these patients.

Therefore, a gut-based therapeutic option that can potentially improve the recurrence rate and the overall prognosis is needed. Fecal transplant has been shown to be effective in conditions with predominant gut-bacterial overgrowth or alteration such as recurrent Clostridium difficile and inflammatory bowel disease. Safe protocols have been developed across the world and studies are being performed in the US under FDA-monitored INDs. Limitations to performing fecal transplant include identifying and screening appropriate donors, which is time consuming and costly, with the cost typically falling to the patient or donor as the required screening is generally not covered by insurance.

The investigators' preliminary data suggest that a one-time administration of an FMT-enema using a rationally-selected donor is safe in patients with cirrhosis and recurrent HE. However, given the small bowel overgrowth and the predominantly small bowel location for bacterial translocation in cirrhosis, which is out of the reach of an enema, an upper GI route for FMT needs to be explored. In the investigators' published experience, a single enema from a rationally-derived donor was associated with significantly lower total and HE-related hospitalizations compared to patients who were randomized to standard of care, with a stable long-term course over >1 year. The investigators' data show that FMT was associated with favorable changes in fecal bile acid (BA) profile with a decrease in proportions of fecal secondary BAs, conjugated BAs and increase in sulfated BAs, indicating a healthier milieu. The investigators also have preliminary data defining the safety of oral FMT capsules in patients with cirrhosis and HE in a current trial led by us. The use of combined oral and rectal routes of FMT, which can potentially alleviate both small bowel and colonic translocation are likely to be better than either alone.

Overall aim: To determine the effect of dual oral and rectal administration of FMT from a rational donor on clinical outcomes (HE and related hospitalizations, brain function, quality of life) and host-microbiota interactions (microbial composition and bile acid composition with systemic and intestinal inflammation), compared to single route of administration and placebo, along with a second oral capsular FMT vs placebo administration in patients with cirrhosis and HE using a randomized, phase II clinical trial.

Design overview: Four groups of outpatients with cirrhosis will be randomized using random sequence generator into placebo and FMT groups and followed for 6 months under an FDA IND double-blind clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosed by either of the following in a patient with chronic liver disease

  * Liver Biopsy
  * Radiologic evidence of varices, cirrhosis or portal hypertension
  * Laboratory evidence of platelet count <100,000 or AST/ALT ratio>1
  * Endoscopic evidence of varices or portal gastropathy
  * Fibroscan values suggestive of cirrhosis
* On treatment for hepatic encephalopathy (patient can be on lactulose and rifaximin)
* Able to give written, informed consent (demonstrated by mini-mental status exam>25 at the time of consenting)
* Women of child bearing potential must agree to use effective contraception for the duration of the study and for 10 days prior and 30 days after the study
* Negative pregnancy test in women of childbearing age

Exclusion Criteria:

* MELD score >22
* WBC count <1000 cells/mm3
* Platelet count<25,000/mm3
* TIPS in place for less than a month
* Currently on antibiotics apart from rifaximin
* Infection at the time of the FMT (diagnosed by blood culture positivity, urinalysis, paracentesis as needed)
* Hospitalization for any non-elective cause within the last 1 month
* Patients who are pregnant or nursing (will be checked using a urine pregnancy test)
* Patients who are incarcerated
* Patients who are incapable of giving their own informed consent
* Patients who are immuno-compromised due to the following reasons:

  * HIV infection (any CD4 count)
  * Inherited/primary immune disorders
  * Current or recent (<3 mos) treatment with anti-neoplastic agent
  * Current or recent (<3 mos) treatment with any immunosuppressant medications [including but not limited to monoclonal antibodies to B and T cells, anti-TNF agents, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine), calcineurin inhibitors (tacrolimus, cyclosporine), mycophenolate mofetil].

    * Subjects who are otherwise immunocompetent and have discontinued any immunosuppressant medications 3 or more months prior to enrollment may be eligible to enroll
* Patients on renal replacement therapy
* Patients with untreated, in-situ colorectal cancer
* Patients with a history of chronic intrinsic GI diseases such as inflammatory bowel disease

  * ulcerative colitis, Crohn's disease or microscopic colitis

    * eosinophilic gastroenteritis or celiac disease
* Major gastro-intestinal or intra-abdominal surgery in the last three months

Other Exclusion Criteria:

* Enema-related

  * Platelet count<25,000
  * Grade IV hemorrhoids
* Safety-related:

  * Dysphagia
  * History of aspiration, gastroparesis, intestinal obstruction
  * Ongoing antibiotic use (except for Rifaximin)
  * Severe anaphylactic food allergy
  * Allergy to ingredients Generally Recognized As Safe in the FMT capsules (glycerol, sodium chloride, hypromellose, gellan gum, titanium dioxide, theobroma oil)
  * Adverse event attributable to prior FMT
  * ASA Class IV or V
  * Pregnant or nursing patients
  * Acute illness or fever within 48 hours of the day of planned FMT
  * Immunocompromised due to medical conditions
  * Probiotics use within the last 48 hours of the day of planned FMT
  * Any condition that the physician investigators deem unsafe, including other conditions or medications that the investigator determines puts the participant at greater risk from FMT

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S. Bajaj, MD MS, Principal Investigator — Hunter Holmes McGuire VA Medical Center, Richmond, VA
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bajaj JS, Fagan A, Sterling RK, Sikaroodi M, Gallagher ML, Lee H, Matherly SC, Bartels A, Mousel T, Davis BC, Puri P, Fuchs M, Thacker LR, McGinley JP, Khoruts A, Gillevet PM. The multi-omic basis for hepatic encephalopathy recurrence: Analysis of the THEMATIC trial. JHEP Rep. 2025 Oct 18;8(1):101634. doi: 10.1016/j.jhepr.2025.101634. eCollection 2026 Jan. PMID 41503571
- [Derived] Bloom PP, Bajaj JS. The Current and Future State of Microbiome Therapeutics in Liver Disease. Am J Gastroenterol. 2024 Jan 1;119(1S):S36-S41. doi: 10.14309/ajg.0000000000002581. No abstract available. PMID 38153225

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with cirrhosis and hepatic encephalopathy
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.5) | 60.6 (10.3) | 63.0 (11.7) | 65.0 (7.1) | 63.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 5 | 12
  Male | 12 | 14 | 12 | 10 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events Related to FMT
Description: Number of patients with serious adverse events between groups related to FMT, especially related to HE
Time Frame: 6 months
Population: number of patients
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Adverse Events Related to FMT
Description: Number of patients with adverse events that do not fit the criteria of serious adverse events between groups related to FMT
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in Microbial Diversity in Stool
Description: Shannon diversity index compared to baseline and engraftment related to the donor at baseline, within 30 days and then monthly till 6 months. Ranges usually from 0-10, higher values represent a better diversity. There are no maximum values.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Number analyzed (Participants) | 15 | 14 | 14 | 14
units on a scale | 1.45 (0.37) | 1.46 (0.33) | 1.71 (0.33) | 1.53 (0.72)

4. Secondary Outcome: Sickness Impact Profile Change
Description: Quality of life assessment change defined by Sickness Impact Profile total score at 30 days and 6 months between groups. This is a percentage result ranges usually from 0-100. A higher score indicates worse quality of life related to the participant's health within 24 hours.
Time Frame: 30 days and 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale | 9.63 [3 to 21] | 15.62 [7.94 to 24.49] | 18.15 [8.78 to 23.59] | 15.94 [13.04 to 26.65]

5. Secondary Outcome: Psychometric Hepatic Encephalopathy Score Performance Change
Description: Cognitive assessment change using the Psychometric hepatic encephalopathy score between groups at 60 days Range is -15 to +5 and higher is better
Time Frame: 60 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Number analyzed (Participants) | 14 | 14 | 14 | 14
score on a scale | -7 [-11 to -3] | -3 [-7 to -2] | -5 [-9 to 1] | -5.5 [-10.25 to 1.75]

6. Secondary Outcome: EncephalApp Stroop Off and On Time Change
Description: Cognitive assessment change using the Stroop Off and On Time change at 60 days and 6 months. This is in seconds. EncephalApp stroop is a computerized test of attention, psychomotor speed and cognitive flexibility. A higher time required to complete 5 correct runs in both Off and On stages is the measure here. There no maximum values but the lower amount of time that is needed, the better is the cognitive function.
Time Frame: 60 days
Measure: Median (Inter-Quartile Range); unit: units on a scale (seconds)
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale (seconds) | 218.5 [175.6 to 281.5] | 194.1 [161.9 to 265.3] | 184.8 [171.1 to 260.0] | 235.3 [177.6 to 248.0]

7. Secondary Outcome: Change in Microbial Diversity in Saliva
Description: Shannon diversity index compared to baseline at 30 days and then monthly till 6 months. Ranges usually from 0-10. Higher values represent a better diversity. There are no maximum values.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Number analyzed (Participants) | 13 | 13 | 12 | 11
units on a scale | 1.55 (0.39) | 1.57 (0.72) | 1.57 (0.30) | 1.56 (0.29)

8. Secondary Outcome: HE Related Events
Description: Number of patients with Hepatic encephalopathy related events
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 6 | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | Group 3: Oral Placebo and Rectal FMT | Group 2: Oral FMT and Rectal Placebo | Group 1: Dual Oral and Rectal FMT
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/15 | 1/15 | 1/15
Serious Adverse Events (participants affected / at risk) | 6/15 | 5/15 | 5/15 | 6/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Group 3: Oral Placebo and Rectal FMT (N=15) | Group 2: Oral FMT and Rectal Placebo (N=15) | Group 1: Dual Oral and Rectal FMT (N=15)
Liver-related hospitalizations (Hepatobiliary disorders) | 6 (9) | 2 (4) | 2 (3) | 2 (4)
Falls (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Seizure recurrence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 3 (4) | 2 (2) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT03796598/Prot_SAP_000.pdf